CLINICAL TRIAL: NCT02350543
Title: Must Aspirin be Discontinued Prior to TURBT: a Prospective, Randomized, Non-inferiority Trial Comparing Peri-operative Aspirin Continuation Versus Discontinuation.
Brief Title: Peri-operative Aspirin Continuation Versus Discontinuation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient recruitment.
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Marc Lubin, Dr., Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMC-13-0666
Record Dates: First submitted 2015-01-26; First posted 2015-01-29 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Hematuria; Urinary Bladder Neoplasms
Keywords: Aspirin usage; Transurethral resection of bladder tumor (TURBT)
MeSH Terms: conditions — Hematuria; Urinary Bladder Neoplasms | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspirin continuation (Active Comparator): Continued use of Acetylsalicylic acid at prior dosage (75mg or 100mg tablet one-per-day).
  Interventions: Drug: Aspirin
- Aspirin discontinuation (No Intervention): Discontinuation of Acetylsalicylic acid ten days prior to surgery, and re-initiation two weeks after hospital discharge.

INTERVENTIONS:
Drug: Aspirin
  Other Names: Acetylsalicylic acid
  Arms: Aspirin continuation

SUMMARY:
This study evaluates the continuation (non-discontinuation) of Aspirin during TURBT. Half of participants will continue their usual low-dose Aspirin regimen during TURBT and throughout the perioperative period, while the other half will discontinue Aspirin use ten days prior to surgery (standard recommendation) and restart therapy two weeks post-discharge.

DETAILED DESCRIPTION:
Recently, the American College of Chest Physicians in their 2012 clinical guidelines on perioperative anti-thrombotic therapy associated TUR of bladder tumour (TURBT) with an increased risk of bleeding associated with anti-thrombotic therapy. Despite this, contemporary series of TURBT identify the rate of significant in-hospital postoperative bleeding at only 2-3.4%. Previous prospective work by our group demonstrated no increase in postoperative hemorrhagic complications with early initiation of Aspirin following TURBT. These findings are supported by a recent retrospective work on TURBT showing a similar complication profile between continued perioperative antiplatelet therapy and antiplatelet naive patients.

The risk associated with Aspirin withdrawal prior to surgery, including increased thrombogenicity, has been extensively studied. Following cessation of Aspirin, full platelet recovery is expected within 12-14 days, however, hemostasis may be regained with as little as 20% of normal platelet activity. Further, evidence supports a platelet rebound phenomenon in the setting of acute Aspirin withdrawal and a resultant clinical prothrombotic state, with thrombotic events peaking ten days following drug cessation. Finally, the acute stress response postoperatively is well known; one component being hypercoagulability which lasts at least seven days after major and uneventful abdominal surgery, predominantly caused by increased platelet activity.

Whereas TURBT generally carries a low overall risk of cardiac morbidity, the general requirement to discontinue Aspirin pre-operatively potentially increases certain patients' cerebrovascular or cardiac risk (eg. post-coronary stent placement). As shown above, the risk of significant post-operative hematuria is minimal, and as such, Aspirin withdrawal may be unnecessary. We will perform a prospective, randomized controlled trial to address the safety and tolerability of continued Aspirin use during TURBT.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 years and older with the ability for self-consent,
* referred for elective TURBT,
* receiving low-dose daily Aspirin prophylaxis.

Exclusion Criteria:

* known coagulopathy or abnormal coagulation profile (prothrombin time, partial thromboplastin time, or platelet count),
* receiving other anti-thrombotic, anti-coagulant, or non-steroidal anti-inflammatory medication (NSAIDs),
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Significant hematuria (composite endpoint) | Post-operative admission period until 45 days post-discharge.
  (Composite endpoint): 1. Requiring bladder catheter drainage (after catheter removal), 2. requiring re-hospitalization, 3. requiring operative intervention (ie. cystoscopy +/- transurethral fulguration). Each sub-element within the composite endpoint will receive a binary score [0,1] to denote occurrence. Similarly, the primary endpoint is a binary measure indicating occurrence of any sub-element. Sub-elements 1-3 (re-cath, re-hospitalization, or cystoscopic intervention) may occur at any point throughout the followup period.

SECONDARY OUTCOMES:
Time to urinary catheter removal | up to 45 days
  Measured in post-operative days, from the time of surgery until catheter removal (typically during post-operative admission period).
Withholding or withdrawal of Aspirin | up to 45 days
  A binary measure [0,1]. In the control group (Aspirin restarted two weeks post-discharge), if Aspirin is withheld due to continued hematuria, this will constitute an event. Similarly, in either group, if Aspirin is withdrawn at any point post-operatively due to hematuria, this will constitute an event.
Time to urine clearance | up to 45 days
  Measured in postoperative days until any lingering, sporadic macrohematuria has resolved. Patients will be discharged with a Hematuria Grading Scale based on that developed by Lee et al, a VAS-like scale of hematuria intensity (redness), and will note their most intense hematuria level on a daily basis until urine clearance. It is assumed that postoperative macrohematuria will resolve by 45 days postoperatively, the duration of followup.

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Lubin, MD, Principal Investigator — Department of Urology, Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- [Background] Douketis JD, Spyropoulos AC, Spencer FA, Mayr M, Jaffer AK, Eckman MH, Dunn AS, Kunz R. Perioperative management of antithrombotic therapy: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e326S-e350S. doi: 10.1378/chest.11-2298. PMID 22315266
- [Background] Nieder AM, Meinbach DS, Kim SS, Soloway MS. Transurethral bladder tumor resection: intraoperative and postoperative complications in a residency setting. J Urol. 2005 Dec;174(6):2307-9. doi: 10.1097/01.ju.0000181797.19395.03. PMID 16280830
- [Background] Collado A, Chechile GE, Salvador J, Vicente J. Early complications of endoscopic treatment for superficial bladder tumors. J Urol. 2000 Nov;164(5):1529-32. PMID 11025697
- [Background] De Nunzio C, Franco G, Cindolo L, Autorino R, Cicione A, Perdona S, Falsaperla M, Gacci M, Leonardo C, Damiano R, De Sio M, Tubaro A. Transuretral resection of the bladder (TURB): analysis of complications using a modified Clavien system in an Italian real life cohort. Eur J Surg Oncol. 2014 Jan;40(1):90-5. doi: 10.1016/j.ejso.2013.11.003. Epub 2013 Nov 12. PMID 24284200
- [Background] Ehrlich Y, Yossepowitch O, Margel D, Lask D, Livne PM, Baniel J. Early initiation of aspirin after prostate and transurethral bladder surgeries is not associated with increased incidence of postoperative bleeding: a prospective, randomized trial. J Urol. 2007 Aug;178(2):524-8; discussion 528. doi: 10.1016/j.juro.2007.03.134. Epub 2007 Jun 14. PMID 17570430
- [Background] Picozzi S, Marenghi C, Ricci C, Bozzini G, Casellato S, Carmignani L. Risks and complications of transurethral resection of bladder tumor among patients taking antiplatelet agents for cardiovascular disease. Surg Endosc. 2014 Jan;28(1):116-21. doi: 10.1007/s00464-013-3136-8. Epub 2013 Sep 4. PMID 24002913
- [Background] Patrignani P, Filabozzi P, Patrono C. Selective cumulative inhibition of platelet thromboxane production by low-dose aspirin in healthy subjects. J Clin Invest. 1982 Jun;69(6):1366-72. doi: 10.1172/jci110576. PMID 7045161
- [Background] Bradlow BA, Chetty N. Dosage frequency for suppression of platelet function by low dose aspirin therapy. Thromb Res. 1982 Jul 1;27(1):99-110. doi: 10.1016/0049-3848(82)90283-3. PMID 7123514
- [Background] Gerstein NS, Schulman PM, Gerstein WH, Petersen TR, Tawil I. Should more patients continue aspirin therapy perioperatively?: clinical impact of aspirin withdrawal syndrome. Ann Surg. 2012 May;255(5):811-9. doi: 10.1097/SLA.0b013e318250504e. PMID 22470078
- [Background] Biondi-Zoccai GG, Lotrionte M, Agostoni P, Abbate A, Fusaro M, Burzotta F, Testa L, Sheiban I, Sangiorgi G. A systematic review and meta-analysis on the hazards of discontinuing or not adhering to aspirin among 50,279 patients at risk for coronary artery disease. Eur Heart J. 2006 Nov;27(22):2667-74. doi: 10.1093/eurheartj/ehl334. Epub 2006 Oct 19. PMID 17053008
- [Background] Mahla E, Lang T, Vicenzi MN, Werkgartner G, Maier R, Probst C, Metzler H. Thromboelastography for monitoring prolonged hypercoagulability after major abdominal surgery. Anesth Analg. 2001 Mar;92(3):572-7. doi: 10.1097/00000539-200103000-00004. PMID 11226080
- [Background] Eagle KA, Berger PB, Calkins H, Chaitman BR, Ewy GA, Fleischmann KE, Fleisher LA, Froehlich JB, Gusberg RJ, Leppo JA, Ryan T, Schlant RC, Winters WL Jr, Gibbons RJ, Antman EM, Alpert JS, Faxon DP, Fuster V, Gregoratos G, Jacobs AK, Hiratzka LF, Russell RO, Smith SC Jr; American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to Update the 1996 Guidelines on Perioperative Cardiovascular Evaluation for Noncardiac Surgery). ACC/AHA guideline update for perioperative cardiovascular evaluation for noncardiac surgery---executive summary a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to Update the 1996 Guidelines on Perioperative Cardiovascular Evaluation for Noncardiac Surgery). Circulation. 2002 Mar 12;105(10):1257-67. No abstract available. PMID 11889023
- [Background] Lee JY, Chang JS, Koo KC, Lee SW, Choi YD, Cho KS. Hematuria grading scale: a new tool for gross hematuria. Urology. 2013 Aug;82(2):284-9. doi: 10.1016/j.urology.2013.04.048. PMID 23896092
- See also: Soni, A. Aspirin use among the adult U.S. non-institutionalized population, with and without indicators of heart disease, 2005. Statistical Brief #179. July 2007. Agency for Healthcare Research and Quality, Rockville, Md. — http://www.meps.ahrq.gov/mepsweb/data_files/publications/st179/stat179.pdf